CLINICAL TRIAL: NCT04293211
Title: Effectiveness of the Adding High Fidelity Simulation to the Bleeding Control
Brief Title: Effectiveness of the Adding High Fidelity Simulation to the Bleeding Control Course in Regards to Proper Tourniquet Placement Amongst School Personnel
Status: Completed | Type: Observational
Sponsor: White Plains Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Stop The Bleed
Record Dates: First submitted 2020-02-25; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Tourniquet Placement; Wound Packing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Upon completion of B-Con presentation, this group will be tested regarding tourniquet placement using the rubric. A tourniquet is regarded as appropriately placed if it is 2 inches above the wound, not located on a joint, appropriate tightness (meaning a finger cannot be placed under it and it is indenting the mannequin). This is as per prior studies. Feedback will be given at the end of this session.
- Simulation: This group will have to interact with a panicked actor/actress as well as the SIM MAN 3G who will have two wounds under his clothes. One that will be actively pumping a large amount of arterial blood that will require tourniquet placement and the other wound with trace venous bleeding that will require simple pressure with a clean cloth. Participants will be given feedback on items that they missed. The observer will fill out the rubric and give feedback to the group.
  Interventions: Other: Simulation

INTERVENTIONS:
Other: Simulation — To measure the efficacy of adding a high-fidelity simulation versus low fidelity simulation to the current B-Con Course. This will be assessed by evaluation of applying tourniquets properly and packing traumatic wounds as well as retention of these skills over a period of time amongst school teachers and security personnel.
  Groups: Simulation

SUMMARY:
This is a joint project by the White Plains School District and White Plains Hospital regarding the training of over 66 school personnel regarding the American College of Surgeons (ACS) "Stop the Bleed" campaign for mass casualty incidents. This project developed from an outreach from White Plains Hospital and an interest from the White Plains School District to work together to train staff in the event of a mass casualty incident / active shooter.

DETAILED DESCRIPTION:
From January through June 2019, participants will be requested to attend one of six sessions that will be held at the hospital simulation center. Participants will be randomized into 1 of 2 study arms. Each participant that enters the B-Con course will be randomized using a "random generator." At the start of the program, all participants will be explained the purpose of the research study and the two groups (Control versus High Fidelity). An option will be given for participants to be able to opt out. So that our participants all have the same opportunities afforded to their colleagues, we will also offer the control group the option to participate in the high fidelity simulation at the conclusion of the entire program.

All groups will sit through the exact same B-Con powerpoint presentation by trained STB instructors. This course includes the powerpoint presentation that reviews how to call for help, assess those affected, identify the location of life-threatening bleed, apply pressure, pack a wound and/or apply a tourniquet and when to do this. Tourniquet placement is taught as is wound packing placement. Participants will each be given tourniquets to practice alongside the instructor. The presentation will cover the first hour of the curriculum. This is considered to be the standard for this course.

Upon conclusion of the course, the control group and high fidelity group will be separated into two rooms based on their randomization. In groups of 2, participants will be trained in tourniquet placement, wound packing. The High Fidelity group will have a simulation intervention in addition and the wound packing will be performed on a device that has biofeedback. Upon conclusion of this one hour session, both groups will be tested on wound packing and tourniquet placement. They will again be tested 3-8 months later on retention for wound packing and tourniquet placement.

ELIGIBILITY:
Inclusion Criteria:

* any volunteer employee who is over the age of 18 that is a staff member at the White Plains School District.

Exclusion Criteria:

* any participants who have prior hemorrhage control training. However, although excluded from the study, they are welcome to participate in the program

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: White Plains School District employees
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Assessment by Evaluation of Applying Tourniquets | 6 months
  Measure correct tourniquet placement based on internally validated scale. Binomial variable (correct or incorrect). Indications for incorrect placement will also be documented (too loose, incorrect location, longer than 7 minutes, participant requested to discontinue).

SECONDARY OUTCOMES:
Assessment by Evaluation of Packing Traumatic Wounds | 6 months
  Amount of pressure placed for 90 seconds using a biofeedback device with a threshold of 25psi based on prior studies on hemorrhage control on porcine models
Retention of Skills Over a Period of Time | 8 months
  Tourniquet and wound packing based on above rubric and biofeedback device, 3-8 months after training
Evaluate the Change in Length of Time to Tourniquet Placement with Simulation Scenario | 6 months
  Measure correct tourniquet placement based on internally validated scale. Binomial variable (correct or incorrect). Indications for incorrect placement will also be documented (too loose, incorrect location, longer than 7 minutes, participant requested to discontinue).

CONTACTS AND LOCATIONS:
Locations (1):
- White Plains Hospital, White Plains, New York, United States

REFERENCES:
- [Derived] Jafri FN, Dadario NB, Kumar A, Silverstein SR, Quintero F, Larsen EA, Fasciglione K, Mirante D, Ellsworth K, Amicucci B, Ricca J. The Addition of High-Technology Into the Stop the Bleed Program Among School Personnel Improves Short-Term Skill Application, Not Long-Term Retention. Simul Healthc. 2021 Dec 1;16(6):e159-e167. doi: 10.1097/SIH.0000000000000546. PMID 33600137